CLINICAL TRIAL: NCT06045039
Title: Clinical Efficacy of Stent-balloon-stent (SBS) Technique in the Treatment of Coronary Bifurcation Lesions
Status: Recruiting | Type: Observational
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Principal Investigator, Xianpei Wang, Chief Physician, Henan Institute of Cardiovascular Epidemiology
Other Study IDs: HenanICE2023
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Coronary Disease; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Myocardial Ischemia
Keywords: Angioplasty; Coronary Angiography; surgery; Coronary Vessels; diagnostic imaging; pathology; Drug-Eluting Stents; Treatment Outcome
MeSH Terms: conditions — Coronary Disease; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Myocardial Ischemia | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stent-balloon-stent (SBS) technique: Patients with coronary bifurcation lesions underwent stent-balloon-stent (SBS) technique. The procedure of this technique is to implant the stent into the side branch at the 1~2mm, which is away from the opening of the branch, and then implant the stent into the main vessel. The guide wire enters the side branch from the mesh at the distal end of the main vascular stent, and the drug balloon is used to dilate the opening of the side branch, so that the opening area of the side branch is more than 5mm².
  Interventions: Other: Stent-balloon-stent (SBS) technique

INTERVENTIONS:
Other: Stent-balloon-stent (SBS) technique — Patients with coronary bifurcation lesions underwent stent-balloon-stent (SBS) technique. The procedure of this technique is to implant the stent into the side branch at the 1~2mm, which is away from the opening of the branch, and then implant the stent into the main vessel. The guide wire enters the side branch from the mesh at the distal end of the main vascular stent, and the drug balloon is used to dilate the opening of the side branch, so that the opening area of the side branch is more than 5mm².

SUMMARY:
The treatment of coronary bifurcation lesions continue to remain challenges. Due to the special hemodynamics caused by the special anatomical structure of the coronary bifurcation, it is easy to cause vascular crest displacement and plaque formation. The existing single-stent strategy and double-stent strategy are easy to cause vascular crest offset, stent accumulation, in-stent thrombosis, in-stent restenosis and other poor long-term prognosis. Stent-balloon-stent (Stent-balloon-stent, SBS) technique enables the guide wire to enter the side branch from the mesh at the distal end of the main vascular stent, and the drug balloon is used to dilate the opening of the side branch, so that the opening area of the side branch is more than 5mm².The SBS technique reduces the risk of branch vascular dissection, occlusion, snow shoveling phenomenon, maintain the original state of bifurcated blood vessels to the greatest extent, should have a good impact on the long-term prognosis of patients with coronary bifurcation lesions (CBL). The purpose of this study is to explore the feasibility, safety and effectiveness of SBS technique.

DETAILED DESCRIPTION:
This is a study to evaluate the application of stent-balloon-stent (Stent-balloon-stent, SBS) in complex bifurcation lesions. 1-2mm from the side branch (SB) opening, the stent was implanted in the side branch, and then the stent was implanted in the main vessel (MV).The guide wire enters the side branch from the mesh at the distal end of the main vascular stent, and the drug balloon is used to dilate the opening of the side branch, so that the opening area of the side branch is more than 5mm².The patients were examined by coronary angiography before operation and 6-12 months after operation, and the related data such as stenosis rate and minimum lumen diameter of diseased vessels were recorded. The incidence of target vessel failure (TLF) 6-12 months later, including cardiogenic death, target vessel myocardial infarction and clinically driven target vessel revascularization, was taken as the main clinical end point. The corresponding data of the patients before and after operation were obtained, and the clinical efficacy was compared with the existing double stent strategy.

ELIGIBILITY:
Inclusion Criteria:

* There is evidence of myocardial ischemia, such as coronary angiography, including patients with stable angina pectoris, unstable angina pectoris, asymptomatic myocardial ischemia and acute myocardial infarction (> 24 hours).
* All bifurcation lesions were Medina 1, 1, 1 or 0, 1, 1 with reference vessel diameter (RVD) in the SB ≥2.5 mm by visual estimation and had to meet DEFINITION criteria of complex bifurcations
* Patients who can tolerate long-term antiplatelet therapy
* None of the vessels related to bifurcation lesions have received stent surgery
* Patients who agree and sign an informed consent form

Exclusion Criteria:

* Patients who are unwilling to sign the relevant informed consent form
* Patients with severe surgical contraindications
* Life expectancy of patients is less than 12 months
* Patients who have previously undergone stent implantation or surgical coronary artery bypass grafting for related lesions
* Patients with severe hepatorenal insufficiency
* Heart failure patients with NYHA grade ≥ Ⅲ
* Patients who are scheduled for surgery requiring antiplatelet medication interruption within 6 months
* Patients who need chronic oral anticoagulation
* Any clinical condition of the patient may interfere with medication compliance or long-term follow-up
* Pregnant or breastfeeding women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had evidence of myocardial ischemia and received interventional therapy for coronary bifurcation lesions in our center from January 2023 to December 2023.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure rate | 3-12 months
  cardiac death
Target lesion failure rate | 6-12 months
  target vessel myocardial infarction (TVMI)
Target lesion failure rate | 6-12 months
  clinically driven target lesion revascularization (TLR)

SECONDARY OUTCOMES:
minimum lumen area and lumen stenosis rate | 6-12months
  minimum lumen area and lumen stenosis rate

CONTACTS AND LOCATIONS:
Overall Officials: Xianpei Wang, MD, Study Chair — FF
Locations (1):
- Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
Others can obtain the individual participant data from the researcher by reasonable request